CLINICAL TRIAL: NCT00323856
Title: Phase IV A Study of Immunologic Safety for Alphanate in Previously Treated Patients Diagnosed With Severe Hemophilia A
Brief Title: Safety Study of Alphanate in Previously Treated Patients With Severe Hemophilia A
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Grifols Biologicals, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GBI 04-01
Record Dates: First submitted 2006-05-08; First posted 2006-05-10 (Estimated); Results first posted 2022-06-09 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Severe Hemophilia A
Keywords: Hemophilia A; Plasma-derived treatment; Factor VIII; Inhibitor
MeSH Terms: conditions — Hemophilia A | interventions — Factor VIII

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Coagulation factor VIII (Human) (Experimental): Anti-Hemophilic coagulation factor VIII (Human) Alphanate SD/HT
  Interventions: Drug: Alphanate SD/HT

INTERVENTIONS:
Drug: Alphanate SD/HT — Plasma-derived preparation of Factor VIII
  Other Names: Anti-hemophilic (human) coagulation factor VIII

SUMMARY:
The purpose of this study is to determine the immunologic and overall safety associated with long-term use of Alphanate in subjects diagnosed with severe hemophilia A (Factor VIII:C less than 0.01 IU/ml), who have been previously treated with plasma-derived Factor VIII products other than Alphanate and who have no history of developing either antibody inhibitors to Factor VIII or nonspecific inhibitors of coagulation.

DETAILED DESCRIPTION:
This is a Phase IV, non-randomized, multicenter study of at least 50 evaluable subjects diagnosed with severe hemophilia A. Enrolled subjects will be treated at home and with in-clinic therapy exclusively with Alphanate as their sole source of Factor VIII concentrate for prophylaxis and treatment of all bleeding episodes and surgical procedures. Subjects will be treated for at least 2 years and a minimum of 50 exposure days, or if 50 exposure days are not reached, for a maximum of 30 months and in accordance with the subject's usual pre-study treatment regimen. Subjects will continue treatment as above or until they develop inhibitors to Factor VIII at a titer greater than or equal to 5 Bethesda units (BU/ml); Factor VIII becomes ineffective at providing hemostasis, or the subject exhibits severe or serious adverse events that prevent completion of the study.

ELIGIBILITY:
Inclusion Criteria:

* Male.
* At least 6 years of age and not more than 65 years of age.
* Signed and dated Informed Consent Form and Patient Authorization for Release of Information approved by the appropriate Institutional Review Board (IRB) prior to screening and enrollment. If the subject is a minor (i.e., less than 18 years of age) both he and his parent or legal guardian must sign and date the informed consent.
* Diagnosis of severe hemophilia A.
* Levels of Factor VIII less than 0.01 IU/mL.
* Treatment with cryoprecipitate, Factor VIII concentrates, and/or whole blood, for at least 150 cumulative exposure days (CEDs) prior to enrollment.
* No treatment with cryoprecipitate, Factor VIII concentrate, or any other blood product, for at least 72 hours prior to screening.
* No previous diagnosis with inhibitors to Factor VIII at any detectable titer.
* Subjects must never have been diagnosed with nonspecific inhibitors of coagulation.
* Negative test for the presence of Factor VIII inhibitors at screening and enrollment.
* CD4 counts greater than or equal to 400 cells/µL.
* Vaccination against hepatitis A and hepatitis B, or evidence of antibodies against hepatitis A and hepatitis B. (A subject who has no prior immunity against hepatitis A will be offered a course of vaccination for hepatitis A).
* Karnofsky Performance Score of at least 50.

Exclusion Criteria:

* Any immunosuppressive medications including intravenous immunoglobulins at the time of enrollment.
* Clinical signs or symptoms of an infection, such as fever, chills or nausea during screening or enrollment.
* History of frequent reactions to Factor VIII concentrates (e.g., chills or headaches).
* Prior treatment with Alphanate® (Solvent-Detergent/ Heat-Treated).
* Immunocompromised (including HIV+ status or has an impaired immune system due to disease or treatment).

Ages: 6 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2003-04-08 (Actual); Primary Completion 2018-12-11 (Actual); Study Completion 2018-12-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Ken Woodward, Study Director — Instituto Grifols SA
Locations (2):
- Poland (2):
  - Oddzial Chorob Wewnetrznych i Hematologii, Poznan, Szkolna
  - Katedra i Klinika Hematologii Collegium Medicum UJ, Krakow

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in Poland at 2 centers from April 8, 2003 to December 14, 2018.
Pre-assignment Details: Male participants diagnosed with severe hemophilia A who have been previously treated with Factor VIII concentrates, cryoprecipitate, or whole blood for a total of 150 cumulative exposure were enrolled. A total of 51 participants were enrolled out of which, 50 participants received the treatment. A total of 45 participants completed the study.
Groups:
- Alphanate: Participants were treated at home and with in-clinic therapy exclusively with Alphanate as their sole source of Factor VIII (FVIII) concentrate for prophylaxis and treatment of all bleeding episodes and surgical procedures for a period of at least two years and a minimum of 50 exposure days, or, if 50 exposure days were not reached, for a maximum of 30 months. An exposure day was defined as any day on which a participant received one or more infusions of any FVIII containing product. Alphanate was administered intravascularly in accordance with the participant's usual pre-study treatment regimen.
Period: Overall Study
Arm/Group | Alphanate
Started | 50
Completed | 45
Not Completed | 5
Not completed — Withdrawal by Subject | 1
Not completed — Was uncooperative and noncompliant | 1
Not completed — Reason not specified | 1
Not completed — Missing | 2

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received at least one infusion of study medication.
Arm/Group | Alphanate
Number analyzed (Participants) | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.8 (14.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 50
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 30
  Hispanic | 8
  Asian | 11
  Other | 1
Subjects with antibody inhibitors to FVIII [Count of Participants; unit: Participants] | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Factor VIII (FVIII) Inhibitor Development
Description: Incidence of FVIII inhibitor development was defined as any result determined positive at a central laboratory (inhibitor titer of greater than 0.6 modified Bethesda Units/milliliters [BU/mL]) using Nijmegen modification of the Bethesda assay.
Time Frame: Up to Month 30
Population: Safety population included all participants who received at least one infusion of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Alphanate
Number analyzed (Participants) | 50
Participants | 0

2. Secondary Outcome: Number of Participants With Adverse Events (AE)
Description: An AE is defined as any untoward medical occurrence in a participant or clinical investigation participant administered a medicinal product or study treatment, and which did not necessarily have a causal relationship with this administration. Here end of study is defined as completion/discontinuation visit.
Time Frame: Up to Month 30
Population: Safety population included all participants who received at least one infusion of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Alphanate
Number analyzed (Participants) | 50
Participants | 30

3. Secondary Outcome: Change From Baseline in Alkaline Phosphatase
Description: The Baseline value was the last non-missing value before study drug was taken and end of study was defined as completion/discontinuation visit. Change from Baseline was calculated by subtracting Baseline value from the post-infusion visit value.
Time Frame: Baseline and Quarterly Visit 1 (Month 3), 2 (Month 6), 3 (Month 9), 4 (Month 12), 5 (Month 15), 6 (Month 18), 7 (Month 21), 8 (Month 24), 9 (Month 27) and 10 (Month 30)
Population: Safety population included all participants who received at least one infusion of study medication. Number analyzed signifies number of participants evaluable at each specified timepoint.
Measure: Mean (Standard Deviation); unit: microkatal per liter (μkat/L)
Arm/Group | Alphanate
Number analyzed (Participants) | 50
microkatal per liter (μkat/L)
  Baseline: number analyzed (Participants) | 44
  Baseline | 2.315 (1.3287)
  Change at Quarterly Visit 1 (Month 3): number analyzed (Participants) | 39
  Change at Quarterly Visit 1 (Month 3) | -0.030 (0.6136)
  Change at Quarterly Visit 2 (Month 6): number analyzed (Participants) | 39
  Change at Quarterly Visit 2 (Month 6) | -0.146 (0.8197)
  Change at Quarterly Visit 3 (Month 9): number analyzed (Participants) | 42
  Change at Quarterly Visit 3 (Month 9) | -0.087 (0.8601)
  Change at Quarterly Visit 4 (Month 12): number analyzed (Participants) | 41
  Change at Quarterly Visit 4 (Month 12) | -0.309 (0.7635)
  Change at Quarterly Visit 5 (Month 15): number analyzed (Participants) | 40
  Change at Quarterly Visit 5 (Month 15) | -0.127 (1.0940)
  Change at Quarterly Visit 6 (Month 18): number analyzed (Participants) | 42
  Change at Quarterly Visit 6 (Month 18) | -0.342 (0.9484)
  Change at Quarterly Visit 7 (Month 21): number analyzed (Participants) | 40
  Change at Quarterly Visit 7 (Month 21) | -0.490 (1.0561)
  Change at Quarterly Visit 8 (Month 24): number analyzed (Participants) | 42
  Change at Quarterly Visit 8 (Month 24) | -0.299 (1.2843)
  Change at Quarterly Visit 9 (Month 27): number analyzed (Participants) | 8
  Change at Quarterly Visit 9 (Month 27) | -1.004 (1.2453)
  Change at Quarterly Visit 10 (Month 30): number analyzed (Participants) | 2
  Change at Quarterly Visit 10 (Month 30) | -0.075 (0.0827)

4. Secondary Outcome: Change From Baseline in Alanine Aminotransferase
Description: as for outcome 3
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: μkat/L
Arm/Group | Alphanate
Number analyzed (Participants) | 50
μkat/L
  Baseline: number analyzed (Participants) | 44
  Baseline | 0.577 (0.6770)
  Change at Quarterly Visit 1 (Month 3): number analyzed (Participants) | 39
  Change at Quarterly Visit 1 (Month 3) | -0.005 (0.2437)
  Change at Quarterly Visit 2 (Month 6): number analyzed (Participants) | 39
  Change at Quarterly Visit 2 (Month 6) | -0.055 (0.2754)
  Change at Quarterly Visit 3 (Month 9): number analyzed (Participants) | 42
  Change at Quarterly Visit 3 (Month 9) | -0.089 (0.3625)
  Change at Quarterly Visit 4 (Month 12): number analyzed (Participants) | 43
  Change at Quarterly Visit 4 (Month 12) | -0.114 (0.4310)
  Change at Quarterly Visit 5 (Month 15): number analyzed (Participants) | 41
  Change at Quarterly Visit 5 (Month 15) | -0.081 (0.3539)
  Change at Quarterly Visit 6 (Month 18): number analyzed (Participants) | 42
  Change at Quarterly Visit 6 (Month 18) | -0.133 (0.4109)
  Change at Quarterly Visit 7 (Month 21): number analyzed (Participants) | 41
  Change at Quarterly Visit 7 (Month 21) | -0.117 (0.3861)
  Change at Quarterly Visit 8 (Month 24): number analyzed (Participants) | 41
  Change at Quarterly Visit 8 (Month 24) | -0.077 (0.3951)
  Change at Quarterly Visit 9 (Month 27): number analyzed (Participants) | 9
  Change at Quarterly Visit 9 (Month 27) | -0.074 (0.1730)
  Change at Quarterly Visit 10 (Month 30): number analyzed (Participants) | 3
  Change at Quarterly Visit 10 (Month 30) | -0.150 (0.2688)

5. Secondary Outcome: Change From Baseline in Aspartate Aminotransferase
Description: as for outcome 3
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: μkat/L
Arm/Group | Alphanate
Number analyzed (Participants) | 50
μkat/L
  Baseline: number analyzed (Participants) | 44
  Baseline | 0.544 (0.6337)
  Change at Quarterly Visit 1 (Month 3): number analyzed (Participants) | 38
  Change at Quarterly Visit 1 (Month 3) | 0.023 (0.1312)
  Change at Quarterly Visit 2 (Month 6): number analyzed (Participants) | 40
  Change at Quarterly Visit 2 (Month 6) | -0.011 (0.2900)
  Change at Quarterly Visit 3 (Month 9): number analyzed (Participants) | 43
  Change at Quarterly Visit 3 (Month 9) | -0.062 (0.3885)
  Change at Quarterly Visit 4 (Month 12): number analyzed (Participants) | 43
  Change at Quarterly Visit 4 (Month 12) | -0.092 (0.4350)
  Change at Quarterly Visit 5 (Month 15): number analyzed (Participants) | 41
  Change at Quarterly Visit 5 (Month 15) | -0.071 (0.3890)
  Change at Quarterly Visit 6 (Month 18): number analyzed (Participants) | 42
  Change at Quarterly Visit 6 (Month 18) | -0.081 (0.4083)
  Change at Quarterly Visit 7 (Month 21): number analyzed (Participants) | 40
  Change at Quarterly Visit 7 (Month 21) | -0.074 (0.3769)
  Change at Quarterly Visit 8 (Month 24): number analyzed (Participants) | 41
  Change at Quarterly Visit 8 (Month 24) | -0.020 (0.3913)
  Change at Quarterly Visit 9 (Month 27): number analyzed (Participants) | 9
  Change at Quarterly Visit 9 (Month 27) | -0.043 (0.0963)
  Change at Quarterly Visit 10 (Month 30): number analyzed (Participants) | 3
  Change at Quarterly Visit 10 (Month 30) | -0.039 (0.0632)

6. Secondary Outcome: Change From Baseline in Lactate Dehydrogenase
Description: as for outcome 3
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: μkat/L
Arm/Group | Alphanate
Number analyzed (Participants) | 50
μkat/L
  Baseline: number analyzed (Participants) | 43
  Baseline | 5.64 (2.089)
  Change at Quarterly Visit 1 (Month 3): number analyzed (Participants) | 40
  Change at Quarterly Visit 1 (Month 3) | -0.07 (0.926)
  Change at Quarterly Visit 2 (Month 6): number analyzed (Participants) | 37
  Change at Quarterly Visit 2 (Month 6) | -0.04 (1.703)
  Change at Quarterly Visit 3 (Month 9): number analyzed (Participants) | 41
  Change at Quarterly Visit 3 (Month 9) | -0.01 (1.595)
  Change at Quarterly Visit 4 (Month 12): number analyzed (Participants) | 40
  Change at Quarterly Visit 4 (Month 12) | -0.31 (2.231)
  Change at Quarterly Visit 5 (Month 15): number analyzed (Participants) | 39
  Change at Quarterly Visit 5 (Month 15) | -0.47 (1.388)
  Change at Quarterly Visit 6 (Month 18): number analyzed (Participants) | 42
  Change at Quarterly Visit 6 (Month 18) | -0.52 (1.814)
  Change at Quarterly Visit 7 (Month 21): number analyzed (Participants) | 40
  Change at Quarterly Visit 7 (Month 21) | -0.65 (1.560)
  Change at Quarterly Visit 8 (Month 24): number analyzed (Participants) | 39
  Change at Quarterly Visit 8 (Month 24) | -0.21 (2.413)
  Change at Quarterly Visit 9 (Month 27): number analyzed (Participants) | 9
  Change at Quarterly Visit 9 (Month 27) | -0.21 (1.497)
  Change at Quarterly Visit 10 (Month 30): number analyzed (Participants) | 3
  Change at Quarterly Visit 10 (Month 30) | 0.22 (0.972)

7. Secondary Outcome: Change From Baseline in Bilirubin
Description: as for outcome 3
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: micromole per liter (μmol/L)
Arm/Group | Alphanate
Number analyzed (Participants) | 50
micromole per liter (μmol/L)
  Baseline: number analyzed (Participants) | 44
  Baseline | 12.346 (6.2515)
  Change at Quarterly Visit 1 (Month 3): number analyzed (Participants) | 40
  Change at Quarterly Visit 1 (Month 3) | 41.387 (255.8005)
  Change at Quarterly Visit 2 (Month 6): number analyzed (Participants) | 40
  Change at Quarterly Visit 2 (Month 6) | -0.815 (5.0952)
  Change at Quarterly Visit 3 (Month 9): number analyzed (Participants) | 42
  Change at Quarterly Visit 3 (Month 9) | 40.485 (253.2611)
  Change at Quarterly Visit 4 (Month 12): number analyzed (Participants) | 43
  Change at Quarterly Visit 4 (Month 12) | 1.461 (7.2030)
  Change at Quarterly Visit 5 (Month 15): number analyzed (Participants) | 41
  Change at Quarterly Visit 5 (Month 15) | -0.031 (4.0146)
  Change at Quarterly Visit 6 (Month 18): number analyzed (Participants) | 41
  Change at Quarterly Visit 6 (Month 18) | 0.759 (4.0038)
  Change at Quarterly Visit 7 (Month 21): number analyzed (Participants) | 40
  Change at Quarterly Visit 7 (Month 21) | 0.498 (5.3277)
  Change at Quarterly Visit 8 (Month 24): number analyzed (Participants) | 42
  Change at Quarterly Visit 8 (Month 24) | 0.060 (4.4453)
  Change at Quarterly Visit 9 (Month 27): number analyzed (Participants) | 8
  Change at Quarterly Visit 9 (Month 27) | 0.760 (2.9257)
  Change at Quarterly Visit 10 (Month 30): number analyzed (Participants) | 3
  Change at Quarterly Visit 10 (Month 30) | -1.539 (3.8664)

8. Secondary Outcome: Change From Baseline in Blood Urea Nitrogen
Description: as for outcome 3
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: millimole per liter (mmol/L)
Arm/Group | Alphanate
Number analyzed (Participants) | 50
millimole per liter (mmol/L)
  Baseline: number analyzed (Participants) | 44
  Baseline | 5.330 (2.8786)
  Change at Quarterly Visit 1 (Month 3): number analyzed (Participants) | 41
  Change at Quarterly Visit 1 (Month 3) | 0.140 (1.8371)
  Change at Quarterly Visit 2 (Month 6): number analyzed (Participants) | 40
  Change at Quarterly Visit 2 (Month 6) | 0.177 (1.8985)
  Change at Quarterly Visit 3 (Month 9): number analyzed (Participants) | 43
  Change at Quarterly Visit 3 (Month 9) | 0.489 (2.1387)
  Change at Quarterly Visit 4 (Month 12): number analyzed (Participants) | 43
  Change at Quarterly Visit 4 (Month 12) | 1.356 (5.6452)
  Change at Quarterly Visit 5 (Month 15): number analyzed (Participants) | 41
  Change at Quarterly Visit 5 (Month 15) | 13.476 (79.9256)
  Change at Quarterly Visit 6 (Month 18): number analyzed (Participants) | 42
  Change at Quarterly Visit 6 (Month 18) | 1.331 (3.6889)
  Change at Quarterly Visit 7 (Month 21): number analyzed (Participants) | 41
  Change at Quarterly Visit 7 (Month 21) | 0.766 (2.2935)
  Change at Quarterly Visit 8 (Month 24): number analyzed (Participants) | 41
  Change at Quarterly Visit 8 (Month 24) | 0.907 (2.7810)
  Change at Quarterly Visit 9 (Month 27): number analyzed (Participants) | 9
  Change at Quarterly Visit 9 (Month 27) | 0.728 (1.4505)
  Change at Quarterly Visit 10 (Month 30): number analyzed (Participants) | 3
  Change at Quarterly Visit 10 (Month 30) | 0.119 (2.0300)

9. Secondary Outcome: Change From Baseline in Creatinine
Description: as for outcome 3
Time Frame: as for outcome 3
Population: Safety population included all participants who received at least one infusion of study medication.Number analyzed signifies number of participants evaluable at each specified timepoint.
Measure: Mean (Standard Deviation); unit: micromole per liter (μmol/L)
Arm/Group | Alphanate
Number analyzed (Participants) | 50
micromole per liter (μmol/L)
  Baseline: number analyzed (Participants) | 44
  Baseline | 61.30 (15.067)
  Change at Quarterly Visit 1 (Month 3): number analyzed (Participants) | 41
  Change at Quarterly Visit 1 (Month 3) | 3.47 (21.125)
  Change at Quarterly Visit 2 (Month 6): number analyzed (Participants) | 40
  Change at Quarterly Visit 2 (Month 6) | -1.76 (12.956)
  Change at Quarterly Visit 3 (Month 9): number analyzed (Participants) | 43
  Change at Quarterly Visit 3 (Month 9) | 4.18 (13.627)
  Change at Quarterly Visit 4 (Month 12): number analyzed (Participants) | 43
  Change at Quarterly Visit 4 (Month 12) | 18.56 (111.453)
  Change at Quarterly Visit 5 (Month 15): number analyzed (Participants) | 41
  Change at Quarterly Visit 5 (Month 15) | 5.80 (18.984)
  Change at Quarterly Visit 6 (Month 18): number analyzed (Participants) | 42
  Change at Quarterly Visit 6 (Month 18) | 5.44 (15.480)
  Change at Quarterly Visit 7 (Month 21): number analyzed (Participants) | 41
  Change at Quarterly Visit 7 (Month 21) | 5.55 (15.475)
  Change at Quarterly Visit 8 (Month 24): number analyzed (Participants) | 42
  Change at Quarterly Visit 8 (Month 24) | 6.11 (18.426)
  Change at Quarterly Visit 9 (Month 27): number analyzed (Participants) | 9
  Change at Quarterly Visit 9 (Month 27) | 4.93 (12.605)
  Change at Quarterly Visit 10 (Month 30): number analyzed (Participants) | 3
  Change at Quarterly Visit 10 (Month 30) | 7.37 (11.367)

10. Secondary Outcome: Number of Participants Human Immunodeficiency Virus Type 1 and 2 (HIV-1/HIV-2), Hepatitis A Virus (HAV), Hepatitis B Virus (HBV), Hepatitis C Virus (HCV) or Parvovirus B19 -Negative at Baseline Who Are Seropositive for Any of These Viruses
Description: Seroconversion based on Enzyme-linked Immunosorbent Assay (ELISA). Seronegative defined as non-reactive in an ELISA test for antibody to the virus in question. Seropositive defined as reactive in an ELISA test for antibody to the virus in question.
Time Frame: Up to Month 30
Population: Safety population included all participants who received at least one infusion of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Alphanate
Number analyzed (Participants) | 50
Participants
  Human Immunodeficiency Virus Type 1 and 2: number analyzed (Participants) | 49
  Human Immunodeficiency Virus Type 1 and 2 | 5
  Hepatitis A Virus: number analyzed (Participants) | 26
  Hepatitis A Virus | 21
  Hepatitis B Virus (HBsAg): number analyzed (Participants) | 46
  Hepatitis B Virus (HBsAg) | 0
  Hepatitis B Virus (HBsAb): number analyzed (Participants) | 8
  Hepatitis B Virus (HBsAb) | 6
  Hepatitis C Virus: number analyzed (Participants) | 28
  Hepatitis C Virus | 3
  Parvovirus B19: number analyzed (Participants) | 13
  Parvovirus B19 | 6

ADVERSE EVENTS:
Time Frame: Up to Month 30
Description: Safety population included all participants who received at least one infusion of study medication.
Arm/Group | Alphanate
All-Cause Mortality (participants affected / at risk) | 0/50
Serious Adverse Events (participants affected / at risk) | 4/50
Other Adverse Events (participants affected / at risk) | 22/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alphanate (N=50)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1
Device Malfunction (General disorders) | 1
Post Procedural Discharge (Injury, poisoning and procedural complications) | 1
Joint Swelling (Musculoskeletal and connective tissue disorders) | 1
Haematuria (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Alphanate (N=50)
Upper Respiratory Tract Infection (Infections and infestations) | 5
Pharyngitis (Infections and infestations) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 8
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 5
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 4
Contusion (Injury, poisoning and procedural complications) | 3
Joint Injury (Injury, poisoning and procedural complications) | 3
Ligament Sprain (Injury, poisoning and procedural complications) | 3
Limb Injury (Injury, poisoning and procedural complications) | 3
Skin Abrasion (Injury, poisoning and procedural complications) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 4
Back Pain (Musculoskeletal and connective tissue disorders) | 3
Pain (General disorders) | 4
Pyrexia (General disorders) | 4
Acne (Skin and subcutaneous tissue disorders) | 3
Haemorrhage (Vascular disorders) | 3
Headche (Nervous system disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Site may publish results from the Study, after providing Sponsor thirty days' notice prior to submitting a manuscript or other materials related to the Study to any outside party. At Sponsors' request, Site will remove any Confidential Information (other than Study results), and Site will upon Sponsors' request, delay publication or presentation for a period of up to one hundred twenty days to allow Sponsor to protect its interests in any Sponsor Inventions.

DOCUMENTS (2):
  • Study Protocol (2007-01-10): https://cdn.clinicaltrials.gov/large-docs/56/NCT00323856/Prot_000.pdf
  • Statistical Analysis Plan (2010-09-29): https://cdn.clinicaltrials.gov/large-docs/56/NCT00323856/SAP_001.pdf